CLINICAL TRIAL: NCT05863819
Title: Effectiveness and Safety of Mobocertinib in Patients With EGFR Exon 20 Insertion NSCLC in Routine Clinical Practice in China: A Prospective, Single-arm, Multicenter, Observational Study
Brief Title: A Real World Study of Mobocertinib in Adults With Lung Cancer in China (MEANING)
Acronym: MEANING-20
Status: Withdrawn | Type: Observational
Why Stopped: Business reason, unrelated to product safety
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-788-4005
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: Drug Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mobocertinib: Participants with EGFR ex20ins positive locally advanced or metastatic NSCLC who have received mobocertinib in China's routine clinical practice setting will be observed in this study. The observation period for each participant is planned to be 18 months, starting from the participant who received mobocertinib enrolled in this study and ending at the earliest occurrence of the completion of 18 months of follow-up, death, loss to follow-up, or withdrawal from the study.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — As this is an observational study, no intervention will be administered in this study.

SUMMARY:
The main aim of this study is to learn about the time from start of mobocertinib to end of treatment with mobocertinib for any reason in Chinese adults with lung cancer who carry a certain gene mutation (epidermial growth factor receptor - EGFR exon 20 insertion mutation) during normal clinical practice.

Participants will be treated with mobocertinib as per their normal routine. Data for this study will be collected from the available medical records of a participant.

DETAILED DESCRIPTION:
This is a non-interventional, prospective, observational study of participants with EGFR ex20ins positive locally advanced or metastatic non-small cell lung cancer (NSCLC) who received mobocertinib in China's routine clinical practice setting. The primary objective of this study is to assess the real-world time-to-treatment discontinuation (rwTTD) of mobocertinib in study participants.

The study will enroll approximately 120 participants. Participants will be enrolled in the following cohort:

• Mobocertinib

Participants will be treated with mobocertinib as per their normal routine treatment. Data for this study will be collected from the available medical records of a participant every 3 months until the end of treatment and follow up (up to 18 months).

This multi-center trial will be conducted in China. The overall duration of the study will be approximately 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with histologically/cytologically confirmed diagnosis of EGFR ex20ins positive locally advanced or metastatic NSCLC by local hospitals.
2. Participants who received mobocertinib as treatment therapy in routine clinical practice; the decision to treat with mobocertinib had to be made independently by physician before enrollment into the study.
3. The decision to treat a participant with mobocertinib had to be made independently by physician before enrollment into the study.

Exclusion Criteria:

1. Participants who are participating in other NSCLC interventional clinical study during the treatment of mobocertinib in this study will be excluded;
2. Other situations that the investigators consider not suitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with EGFR ex20ins positive locally advanced or metastatic NSCLC who have received mobocertinib in China's routine clinical practice setting.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-03-30 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Real-World Time-to-Treatment Discontinuation (rwTTD) | Up to 18 months
  Real-world time-to-treatment discontinuation (rwTTD) is defined as the time from initiation of mobocertinib to discontinuation of treatment with mobocertinib for any reason, including disease progression, death, serious adverse events, or participant preference.

SECONDARY OUTCOMES:
Real-World Overall Response Rate (rwORR) | Up to 18 months
  rwORR is defined as the percentage of participants who are confirmed to achieved complete response (CR) or partial response (PR) after receiving mobocertinib in a real word setting. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. CR is defined as disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm.
Real-World Duration of Response (rwDOR) | Up to 18 months
  rwDOR is defined as the time from the measurement criteria are first met for CR/PR (whichever is first recorded) for participants who have achieved confirmed objective response rate (ORR) after receiving mobocertinib to progression or death in a real word setting.
Real-World Disease Control Rate (rwDCR) | Up to 18 months
  rwDCR is defined as the percentage of participants who are confirmed to achieved CR or partial response PR or stable disease (SD) after receiving mobocertinib in a real word setting.PR: partial reduction in size of visible disease in some, or all, areas without any increase in visible disease. SD: no change in overall size of visible disease, or mixed response (some lesions increased, some lesions decreased).
Median Real-World Progression-Free Survival (rwPFS) | Up to 18 months
  rwPFS is defined as the time from initiation of mobocertinib to disease progression or death from any cause, or the time of the last confirmed survival in real world setting.
Real-World PFS (rwPFS) Rate at 1-year, 1.5-year and 2-year | Up to 2 years
  rwPFS rate at 1-year, 1.5-year and 2-years are defined as the probability of progression free survival over one year from initiation of mobocertinib and the probability of progression-free survival over 1.5 years from initiation of mobocertinib. If data is available, the probability of progression-free survival over 2 years from initiation of mobocertinib will also be calculated.
Real-World Overall Survival (rwOS) Rate at 1-year, 1.5-year and 2-year | Up to 2 years
  rwOS rate at 1-year, 1.5-year, and 2-year are defined as the probability of overall survival over one year from initiation of mobocertinib and the probability of overall survival over 1.5 years from initiation of mobocertinib. If data is available, the probability of overall survival over 2 years from initiation of mobocertinib will also be calculated.
Time to Deterioration (TTD) Based on Physical Functioning per European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30) (v3.0) Scale | Up to 18 months
  TTD is defined as the time from baseline to the occurrence of first clinical meaningful deterioration compared to baseline score of EORTC QLQ-C30. TTD will be assessed using QLQ-30 physical function scale using the Kaplan-Meier Method.
TTD Based on Cough per EORTC Quality of Life Questionnaire Lung Cancer module (QLQ-LC13) Scale | Up to 18 months
  TTD is defined as the time from baseline to the occurrence of first clinical meaningful deterioration compared to baseline score of EORTC QLQ-LC13. TTD will be assessed using QLQ-LC13 cough scale using the Kaplan-Meier Method.
TTD Based on Dyspnea per EORTC QLQ-LC13 Scale | Up to 18 months
  TTD is defined as the time from baseline to the occurrence of first clinical meaningful deterioration compared to baseline score of EORTC QLQ-LC13. TTD will be assessed using QLQ-LC13 dyspnea scale using the Kaplan-Meier Method.
TTD Based on Chest Pain Scores per EORTC QLQ-LC13 Scale | Up to 18 months
  TTD is defined as the time from baseline to the occurrence of first clinical meaningful deterioration compared to baseline score of EORTC QLQ-LC13. TTD will be assessed using QLQ-LC13 chest pain scores using the Kaplan-Meier Method.
Number of Participants Categorized with Demographic Characteristics at Baseline | At Baseline (Day 1)
  Demographic characteristics will include age, gender, smoking history, smoking status and family history for malignancies.
Number of Participants Categorized with Clinicopathological Characteristics at Baseline | At Baseline (Day 1)
  Clinicopathological characteristics will include Eastern Cooperative Oncology Group Performance Status (ECOG PS); medical history including clinically significant disease, surgeries, cancer history; current status of lung cancer; comorbidity; Histology: adenocarcinoma, squamous cell carcinoma, mixed, or others; EGFR mutation testing; and co-mutation status.
Number of Participants Categorized with Co-Mutation Characteristics at Baseline | At Baseline (Day 1) at the timing of mobocertinib initiation date
  Co-Mutation characteristics will include gene mutation testing methods and results in participants.
Number of Participants with Adverse Events (AEs) Related to Mobocertinib | Up to 18 months
  AEs refer to any reasons leading to the dose modification, interruption or discontinuation of mobocertinib in Chinese participants with EGFR ex20ins positive locally advanced or metastatic NSCLC in real world setting. Data will be collected from the participant's medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Shanghai Lung Cancer Center, Shanghai Chest Hospital, Shanghai Jiaotong University, P. R. China, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/73db6ead051540ab?idFilter=%5B%22TAK-788-4005%22%5D